CLINICAL TRIAL: NCT01705106
Title: A Drug-drug Interaction Study of Capecitabine and Celecoxib in Patients With Advanced Solid Malignancies
Brief Title: Capecitabine and Celecoxib in Patients With Solid Cancers That Have Been Previously Treated With Standard Therapies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated early due to slow accrual.
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-1318; NCI-2012-01704 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-10-08; First posted 2012-10-12 (Estimated); Results first posted 2018-05-30 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-04

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — Capecitabine; Celecoxib; Pharmacogenomic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (capecitabine, celecoxib) (Experimental): Patients receive celecoxib PO BID for 7 days (course 0) and then on days 1-21 of course 1 and all subsequent courses. Patients also receive capecitabine PO BID on days 1-14 beginning in course 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: capecitabine; Drug: celecoxib; Other: pharmacological study; Other: laboratory biomarker analysis; Other: pharmacogenomic studies

INTERVENTIONS:
Drug: capecitabine — Given PO
  Other Names: CAPE; Ro 09-1978/000; Xeloda
Drug: celecoxib — Given PO
  Other Names: Celebrex; SC-58635
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacogenomic studies — Correlative studies
  Other Names: Pharmacogenomic Study

SUMMARY:
This clinical trial studies capecitabine and celecoxib in treating patients with solid malignancies that are metastatic or cannot be removed by surgery. Drugs used in chemotherapy, such as capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Celecoxib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving capecitabine and celecoxib together may be an effective treatment for solid malignancies.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare steady state pharmacokinetics (PK) (primarily minimum concentration [Cmin], maximum concentration [Cmax], and area under the curve [AUC]) of celecoxib on day 7 of monotherapy versus on day 14 of concomitant administration with capecitabine.

SECONDARY OBJECTIVES:

I. To develop a celecoxib PK drug interaction model using longitudinal data and determine whether the results are concordant with results from the primary objective.

II. To assess the impact of known cytochrome P450 2C9 (CYP2C9) pharmacogenetic variants with reduced enzyme activity (CYP2C9*2 and *3) on the between subject variability in celecoxib PK.

III. To assess tumor response by the Response Evaluation Criteria In Solid Tumors (RECIST, version 1.1) and explore whether there is any correlation between celecoxib PK and response.

IV. To assess toxicity by the Common Terminology Criteria for Adverse Events (CTCAE, version 4.0) and explore whether there is any correlation between celecoxib PK and toxicities related to either celecoxib or capecitabine.

OUTLINE:

Patients receive celecoxib orally (PO) twice daily (BID) for 7 days (course 0) and then on days 1-21 of course 1 and all subsequent courses. Patients also receive capecitabine PO BID on days 1-14 beginning in course 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed solid tumor that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective

OR

Histologically or cytologically confirmed solid tumor for which single agent capecitabine is an appropriate treatment option.

* Eastern Cooperative Oncology Group (ECOG) performance status =< 1
* Life expectancy > 3 months
* Absolute neutrophil count (ANC) >= l500/ul
* Hemoglobin >= 9g/dL
* Platelets >= 100,000/ul
* Creatinine within institutional normal limits or glomerular filtration rate >= 50 mL/min/1.73 m^2 by Chronic Kidney Disease Epidemiology Collaboration (CKD EPI) equation
* Total bilirubin < 1.5 x upper limit of normal
* Serum glutamic oxaloacetic transaminase (SGOT) and serum glutamic pyruvate transaminase (SGPT) < 2.5 x upper limit of normal for patients without liver metastases OR SGOT and SGPT < 5 x upper limit of normal for patients with liver metastases
* Measurable or non-measurable disease will be allowed
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation, up until 30 days after final study treatment; should a woman become pregnant or suspect that she is pregnant while participating in this study, she should inform her treating physician immediately
* Patients taking substrates of CYP2C9 should be encouraged to switch to alternative drugs whenever possible, given the potential for drug-drug interactions with the study drugs
* Signed informed consent

Exclusion Criteria:

* Prior treatment with capecitabine and/or celecoxib is allowed; however, patients with a documented history (at the time of enrollment) of >= grade 3 toxicities with capecitabine or celecoxib are excluded
* Patients taking any of the following drugs are excluded: inducers or inhibitors of CYP2C9, warfarin, aspirin, corticosteroids, or non-steroidal anti-inflammatory drugs (NSAIDs)
* History of myocardial infarction or stroke within the last 6 months, or history of uncontrolled cardiovascular or cerebrovascular disease; a 12-lead electrocardiogram (ECG) will be performed during the screening period
* History of perforation or bleeding related to peptic ulcer disease
* History of hypersensitivity or allergy to study drugs, aspirin, sulfonamides, or NSAIDs
* Known poor metabolizers of CYP2C9 substrates
* Known deficiency of dihydropyrimidine dehydrogenase (DPD)
* Patients who have had chemotherapy, immunotherapy, or investigational anti-cancer therapy within 4 weeks of starting study drug, or radiotherapy within 14 days of starting study drug, or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients may not be receiving any other investigational agents or any concomitant antineoplastic therapy, with the exception of androgen ablating agents (for patients with prior prostate cancer)
* Serious underlying medical or psychiatric illnesses that would, in the opinion of the treating physician, substantially increase the risk for complications related to treatment; similarly, any unstable medical condition that in the opinion of the treating physician or study investigators, would interfere with determination of the study objectives
* Pregnancy or breastfeeding
* Major surgery within 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2012-08-29 (Actual); Primary Completion 2016-02-10 (Actual); Study Completion 2016-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manish R. Sharma, M.D., Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (1):
- University of Chicago Comprehensive Cancer Center, Chicago, Illinois, United States

REFERENCES:
- [Derived] Wood K, Byron E, Janisch L, Salgia R, Sharma MR. Capecitabine and Celecoxib as a Promising Therapy for Thymic Neoplasms. Am J Clin Oncol. 2018 Oct;41(10):963-966. doi: 10.1097/COC.0000000000000400. PMID 28654574

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Capecitabine, Celecoxib)
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Capecitabine, Celecoxib)
Number analyzed (Participants) | 21
Age, Continuous [Median (Full Range); unit: years] | 57.5 [52 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: AUC of Celecoxib on Combination Therapy (Day 14) and AUC of Celecoxib on Celecoxib Monotherapy(Day 7)
Description: These parameters will be estimated for each subject under each treatment condition. The mean ratios (combination therapy/celecoxib monotherapy) will then be estimated together with 90% confidence intervals (CI).
Time Frame: Day 7 and 14 post treatment
Population: The study was terminated early due to slow accrual, thus none of participants was analyzed. Data were not collected.
Arm/Group | Treatment (Capecitabine, Celecoxib)
Number analyzed (Participants) | 0

2. Secondary Outcome: CYP2C9 Genotype
Description: Polymorphisms *2 and *3 will be genotyped and analyzed for their impact on celecoxib AUC using analysis of variance (ANOVA), controlling for gender, age, and other covariates.
Time Frame: one week
Population: The study was terminated early due to slow accrual, thus none of participants was analyzed. Data were not collected.
Arm/Group | Treatment (Capecitabine, Celecoxib)
Number analyzed (Participants) | 0

3. Secondary Outcome: Response Rate
Description: Logistic regression analysis will be performed to describe the relationship (if any) between celecoxib AUC and response rate.
Time Frame: Up to 2 years
Population: The study was terminated early due to slow accrual, thus none of participants was analyzed. Data were not collected.
Arm/Group | Treatment (Capecitabine, Celecoxib)
Number analyzed (Participants) | 0

4. Secondary Outcome: Drug-related Toxicities
Description: Ordinal logistic regression modeling will be used to explore the relationship between celecoxib AUC and toxicity.
Time Frame: Up to six months
Population: The study was terminated early due to slow accrual, thus none of participants was analyzed. Data were not collected.
Arm/Group | Treatment (Capecitabine, Celecoxib)
Number analyzed (Participants) | 0

5. Secondary Outcome: PK Drug Interaction Model
Description: NONMEM software will be used to develop a model describing the drug interaction between capecitabine and celecoxib using PK data collected during the first four weeks of the study.
Time Frame: 4 weeks
Population: The study was terminated early due to slow accrual, thus none of participants was analyzed. Data were not collected.
Arm/Group | Treatment (Capecitabine, Celecoxib)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Patients were followed for 30 days post treatment.
Arm/Group | Treatment (Capecitabine, Celecoxib)
Serious Adverse Events (participants affected / at risk) | 9/21
Other Adverse Events (participants affected / at risk) | 20/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Capecitabine, Celecoxib) (N=21)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1
Chest pain (Cardiac disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other (Pneumonia) (Respiratory, thoracic and mediastinal disorders) | 2
Seizure (Nervous system disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Capecitabine, Celecoxib) (N=21)
Abdominal Pain (Gastrointestinal disorders) | 5
Agitation (Psychiatric disorders) | 1
Anal hemorrhage (Gastrointestinal disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 9
Back pain (Musculoskeletal and connective tissue disorders) | 1
Blood bilirubin increased, intermittent (Gilbert's syndrome) (Investigations) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Bullous dermatitis (on heels from treadmill) (Skin and subcutaneous tissue disorders) | 1
Cataract, right eye (Eye disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Creatinine increased (Investigations) | 1
Diarrhea (Gastrointestinal disorders) | 11
Dizziness (Nervous system disorders) | 2
Dry skin, palms (Skin and subcutaneous tissue disorders) | 1
Dysgeusia (Nervous system disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7
Eye infection, left eye staph infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Fatigue (General disorders) | 12
Fever (General disorders) | 1
Flank pain, right (Musculoskeletal and connective tissue disorders) | 1
Gastrointestinal disorders - Other (Excessive saliva) (Gastrointestinal disorders) | 1
Headache, intermittent (Nervous system disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Hot flashes (Vascular disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hypertension (Vascular disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypotension, orthostatic (Vascular disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Infections and infestations - Other (Black thrush) (Infections and infestations) | 1
Infections and infestations - Other (Oral thrush) (Infections and infestations) | 1
Infections and infestations - Other (Right hand laceration) (Infections and infestations) | 1
Injury, poisoning and procedural complications - Other (Pulled posterior left chest wall muscle) (Injury, poisoning and procedural complications) | 1
Insomnia (Psychiatric disorders) | 3
Lip infection, herpes skin lesion upper lip (Infections and infestations) | 1
Lip pain (Gastrointestinal disorders) | 1
Mucositis (Gastrointestinal disorders) | 4
Mucositis oral (Gastrointestinal disorders) | 2
Nail infection (Infections and infestations) | 1
Nausea (Gastrointestinal disorders) | 8
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Neutrophil count decreased (Investigations) | 1
Non-cardiac chest pain (General disorders) | 1
Oral dysesthesia, intermittent (Gastrointestinal disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Pain, intermittent left sided pain (General disorders) | 1
Pain, left shoulder (General disorders) | 1
Pain, Right shoulder pain (General disorders) | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 12
Papulopustular rash, hands (Infections and infestations) | 1
Paresthesia, right arm (Nervous system disorders) | 1
Paresthesia, Right eye over cheek (Nervous system disorders) | 1
Paronychia (Infections and infestations) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 4
Platelet count decreased (Investigations) | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Postnasal drip, intermittent (Respiratory, thoracic and mediastinal disorders) | 2
Proctitis (Gastrointestinal disorders) | 1
Psychiatric disorders - Other (rage/altered mental status) (Psychiatric disorders) | 1
Rash, back and hands (Skin and subcutaneous tissue disorders) | 1
Rash, forearms (Skin and subcutaneous tissue disorders) | 1
Rash, scrotum (Skin and subcutaneous tissue disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other (Pneumonia) (Respiratory, thoracic and mediastinal disorders) | 2
Skin and subcutaneous tissue disorders - Other (hypochromic lesions chest/nipples) (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other (Night sweats) (Skin and subcutaneous tissue disorders) | 1
"Skin and subcutaneous tissue disorders - Other (Skin lesion right shoulder)" (Skin and subcutaneous tissue disorders) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Stomach pain (Gastrointestinal disorders) | 1
Tachycardia (Cardiac disorders) | 1
Thromboembolic event (pulmonary embolism) (Surgical and medical procedures) | 1
Tremor, hands (Nervous system disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Vomiting (Gastrointestinal disorders) | 4
Weight loss (Investigations) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No